CLINICAL TRIAL: NCT04569162
Title: Rhizomelic Chondrodysplasia Punctata Registry at Nemours Children's Health
Brief Title: Rhizomelic Chondrodysplasia Punctata Registry
Status: Recruiting | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: RhizoKids International (Unknown)
Responsible Party: Principal Investigator, Mahim Jain, Physician, Nemours Children's Clinic
Other Study IDs: MB002
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: RCDP - Rhizomelic Chondrodysplasia Punctata; RCDP1; RCDP2; RCDP3; RCDP4; RCDP5
MeSH Terms: conditions — Chondrodysplasia Punctata, Rhizomelic; Rhizomelic chondrodysplasia punctata, type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this registry is to collect medical information on individuals with rhizomelic chondrodysplasia punctata and closely related conditions. The study team hopes to learn more about these conditions and improve the care of people with it by establishing this registry.

DETAILED DESCRIPTION:
The goal of this registry is to collect information on individuals with rhizomelic chondrodysplasia punctata (also called RCDP). This registry will enable detailed natural history studies of RCDP, with the hopes that identification of risk factors will allow for preventative treatments and thus a better quality of life for individuals with these diagnoses.

This study is limited to chart review, after signed informed consent obtained. There will be no additional visits or time in clinic because of participation in this registry. This study involves only the collection and storage of data extracted from the medical record. Records that may be requested and reviewed as a part of this study include but may not be limited to: specialist evaluations, surgical reports, results of blood and urine tests, genetic testing, x-rays, CT/MRI imaging. There are no special procedures, visits, or expectations of the individual as a result of participation in this registry. No one will be asked to have any specific testing for the sole purposes of this research.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RCDP or closely related conditions by metabolic and/or genetic testing

Exclusion Criteria:

* Not meeting diagnosis of RCDP or closely related conditions by study team physician review of prior metabolic and/or genetic testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any individual at any age with rhizomelic chondrodysplasia punctata or a closely related condition
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05-17 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Characterizations of the natural history of rhizomelic chondrodysplasia punctata | 5 years
  Data will be collected at enrollment, and over time, to allow for analysis of associated features throughout the lifespan
Identification of clinical features that are predictive of poor outcomes | 5 years
  Identifying risk factors will allow for preventative treatments and thus a better quality of life for individuals with RCDP.

CONTACTS AND LOCATIONS:
Overall Officials: Mahim Jain, MD, PhD, Principal Investigator — Nemours
Locations (1):
- Nemours, Wilmington, Delaware, United States